CLINICAL TRIAL: NCT01692743
Title: Telemedicine in Patients With Inflammatory Bowel Disease (TELE-IBD)
Acronym: TELE-IBD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Pittsburgh (Other); Vanderbilt University (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Raymond Cross, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HP-00049230
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis
Keywords: Telemedicine; Inflammatory bowel disease; Crohn's disease; Ulcerative colitis; Quality of life; Health care utilization
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Patient Acceptance of Health Care | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of Care (No Intervention): Participants undergo usual follow up (routine and as needed office visits and telephone calls) and receive educational fact sheets from the Crohn's and Colitis Foundation of America.
- Weekly Home Monitoring (Experimental): Participants log onto the TELE-IBD website weekly to answer questions about disease symptoms, adherence, side effects, to check body weight and to receive educational content. Participants receive self action plans after each self-testing session. Alerts are generated to the nurse coordinator if certain clinical criteria are met.
  Interventions: Behavioral: Home Monitoring
- Home Monitoring Every Other Week (Experimental): Participants log onto the TELE-IBD website every other week to answer questions about disease symptoms, adherence, side effects, to check body weight and to receive educational content. Participants receive self action plans after each self-testing session. Alerts are generated to the nurse coordinator if certain clinical criteria are met.
  Interventions: Behavioral: Home Monitoring

INTERVENTIONS:
Behavioral: Home Monitoring — Participants log onto the TELE-IBD website weekly to answer questions about disease symptoms, adherence, side effects, to check body weight and to receive educational content. Participants receive self action plans after each self-testing session. Alerts are generated to the nurse coordinator if certain clinical criteria are met.
  Arms: Weekly Home Monitoring
Behavioral: Home Monitoring — Participants log onto the TELE-IBD website every other week to answer questions about disease symptoms, adherence, side effects, to check body weight and to receive educational content. Participants receive self action plans after each self-testing session. Alerts are generated to the nurse coordinator if certain clinical criteria are met.
  Arms: Home Monitoring Every Other Week

SUMMARY:
Improved methods are needed to monitor patients with inflammatory bowel disease. Telemedicine has shown promise in patients with other chronic diseases; pilot testing in our patients with inflammatory bowel disease demonstrated that the technology was feasible and improved clinical outcomes.

The telemedicine system for patients with inflammatory bowel disease (Tele-IBD) should improve outcomes for patients, improve access to care in areas with limited resources, and decrease health care costs.

DETAILED DESCRIPTION:
Introduction: Inflammatory bowel disease (IBD) is a chronic condition that results in debilitating symptoms. Although effective treatments exist, inadequate monitoring of symptoms and side effects, nonadherence, and poor patient knowledge are barriers to success. Telemedicine has been used in other chronic diseases to improve outcomes; pilot testing of telemedicine demonstrated that it is feasible and accepted in IBD. Our preliminary results from a randomized trial in participants with ulcerative colitis showed significant improvements in quality of life from baseline to one year in the telemanagement group.

Study Design: Telemedicine for Patients with Inflammatory Bowel Disease (Tele-IBD) is a 12-month, multicenter, randomized, controlled trial to assess the impact of Tele-IBD compared to standard care in participants with IBD. The aims of the study are to: (1) assess disease activity in participants with IBD using Tele-IBD compared to participants using standard care, (2) assess quality of life in participants with IBD using Tele-IBD compared to participants using standard care, and (3) estimate differences of person-level rates of utilization of health care resources in participants with IBD using Tele-IBD compared to participants using standard care.

Methods: Tele-IBD consists of a web-portal and a weight scale. Participants answer questions about IBD symptoms, side effects and adherence using their home PC or a laptop with wireless Internet access provided to them for the study. A series of educational topics is administered via video messaging every 2-3 weeks. Tele-IBD participants complete self-testing weekly or every other week; the results are immediately available on the web-portal for review. Based on the responses, alerts and action plans are created for each participant. A nurse care coordinator consults the participant's medical provider for management changes if necessary. IBD patients evaluated at the University of Maryland, Baltimore, University of Pittsburgh, and Vanderbilt University will be invited to participate. Interested patients will be randomized in a 1:1:1 fashion to receive Tele-IBD weekly, Tele-IBD every other week, or standard care. Disease activity, quality of life, medical adherence, and utilization of health care resources will be assessed every 6 months for one year. In addition, provider interactions with patients in all three arms will be monitored and recorded.

Expected Findings: Tele-IBD will decrease disease activity and improve quality of life through improved adherence and monitoring of symptoms, earlier and more effective implementation of therapy, more frequent patient-provider interactions, and improved patient self-management. Better control of IBD will result in decreased utilization of health care resources.

Significance: If Tele-IBD improves outcomes, it is likely to be used to improve IBD care, to contain health care costs, to increase access to care, and to improve adherence with physician performance measures.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's disease, ulcerative colitis or indeterminate colitis

Exclusion Criteria:

* Cannot comprehend simple instructions in English
* Inability to comply with the study protocol (i.e., active drug or alcohol abuse or history of nonadherence to medical visits and/or medications)
* Presence of an ileostomy, colostomy, ileoanal j pouch anastomosis or ileorectal anastomosis
* Imminent surgery
* History of short bowel syndrome
* No flares of disease in last two years
* Uncontrolled medical or psychiatric disease Degenerative neurologic condition Unstable angina Class III/IV congestive heart failure Severe asthma or chronic obstructive pulmonary disease Symptomatic peripheral vascular disease Chronic renal insufficiency (creatinine > 2.0) Malignancy within the last 5 years (excluding squamous or basal cell cancers of the skin) Poorly controlled depression, mania, and schizophrenia Active infection Acquired immunodeficiency syndrome
* Pregnancy
* Age less than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond K Cross, MD, MS, AGAF, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Cross RK, Jambaulikar G, Langenberg P, Tracy JK, Collins JF, Katz J, Regueiro M, Schwartz DA, Quinn CC. TELEmedicine for Patients with Inflammatory Bowel Disease (TELE-IBD): Design and implementation of randomized clinical trial. Contemp Clin Trials. 2015 May;42:132-44. doi: 10.1016/j.cct.2015.03.006. Epub 2015 Mar 24. PMID 25812483

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Weekly Home Monitoring | Home Monitoring Every Other Week
Started | 117 | 116 | 115
Completed | 90 | 81 | 88
Not Completed | 27 | 35 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Weekly Home Monitoring | Home Monitoring Every Other Week | Total
Number analyzed (Participants) | 117 | 116 | 115 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.7) | 36.4 (11.5) | 40.1 (13.2) | 38.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 66 | 67 | 197
  Male | 53 | 50 | 48 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 116 | 115 | 113 | 344
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 5 | 5 | 24
  White | 100 | 111 | 108 | 319
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 1 | 4
Quality of Life (IBDQ) [Mean (Standard Deviation); unit: units on a scale] — The Inflammatory Bowel Disease Questionnaire (IBDQ) score ranges from 32-224, with higher scores indicating greater disease-specific quality of life. An IBDQ score of greater than 168 has been shown to correlate with clinical remission in patients with Crohn's disease. Further, scores of 16 to 32 have been found to be significant changes when compared to baseline values.
  units on a scale | 168.1 (34) | 172.3 (34.5) | 172.3 (33.1) | 171.0 (33.8)

OUTCOME MEASURES:

1. Primary Outcome: Harvey Bradshaw Index
Description: Disease activity measure for patients with Crohn's disease. The activity index is comprised of 5 items. General well being (0-4), abdominal pain (0-3), number of liquid stools per day (no maximum score), presence of an abdominal mass on physical exam (0-3), and complications (1 point per item). The total score is the sum of the individual parameters with scores less than 5 consistent with clinical remission. The minimum score is 0 and there is no pre-specified maximum score as it depends on the number of liquids stools.
Time Frame: 12 months
Population: Crohn's disease population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Weekly Home Monitoring | Home Monitoring Every Other Week
Number analyzed (Participants) | 79 | 78 | 79
units on a scale | 3.7 (3.6) | 3.2 (3.4) | 4.2 (3.9)

2. Primary Outcome: Inflammatory Bowel Disease Questionnaire
Description: Description: A quality of life (QoL) questionnaire for patients with inflammatory bowel diseases [1].
  Format: 32 questions grouped into four dimensions: bowel, systemic, social, and emotional.
  Scoring: Scores for each question range from 1 (poorest QoL) to 7 (best QoL). The overall range for the 32 item questionnaire is 32-224 with higher scores indicate better QoL. Scores >168 have been shown to correlate with clinical remission in patients with Crohn's disease and a change in score of 16-32 points is considered significant.
Time Frame: 12 months
Population: IBDQ Scores
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Weekly Home Monitoring | Home Monitoring Every Other Week
Number analyzed (Participants) | 117 | 116 | 115
units on a scale | 179.3 (28.2) | 179.2 (32.8) | 181.5 (28.2)

3. Secondary Outcome: Health Care Utilization
Description: Total healthcare encounters 1 year post randomization (a specific scale was not used, simple counts of all encounters after randomization were carried out)
Time Frame: One year
Measure: Number; unit: Encounters
Arm/Group | Standard of Care | Weekly Home Monitoring | Home Monitoring Every Other Week
Number analyzed (Participants) | 117 | 116 | 115
Encounters | 2435 | 2167 | 2481

ADVERSE EVENTS:
Arm/Group | Standard of Care | Weekly Home Monitoring | Home Monitoring Every Other Week
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/116 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/116 | 0/115
Other Adverse Events (participants affected / at risk) | 0/117 | 0/116 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No